CLINICAL TRIAL: NCT06740643
Title: Evaluation of Intracanal Reinforcement with Short Composite Post in Upper Primary Incisors: Randomized Clinical Trial
Brief Title: Evaluation of Intracanal Reinforcement with Short Composite Post in Upper Primary Incisors with Severly Carious Teeth As in Early Childhood Caries Cases Using Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Osama Abdelazeem, master's student at Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: intracanal reinforcement
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Composite Post; Intracanal Reinfocement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intracanal reinforcement with short compsite post (Experimental)
  Interventions: Procedure: intracanal reinforcement using short composite post
- no intracanal reinforcement (Active Comparator)
  Interventions: Procedure: no intracanal reinforcement

INTERVENTIONS:
Procedure: intracanal reinforcement using short composite post — after pupectomy is done flowable composite will be applied 3mm intacanal to make a short compsite post before zircon crown aplicaction
  Arms: intracanal reinforcement with short compsite post
Procedure: no intracanal reinforcement — no intracanal reinforcement using resin modified glass ionmer before zircon crown application
  Arms: no intracanal reinforcement

SUMMARY:
Severely damaged incisors may lead to difficulty in speech, decreased masticatory efficiency, abnormal tongue habits, subsequent malocclusions, and psychological and self-esteem problems. There are several methods mentioned in the literature for the restoration of severely decayed primary anterior teeth. The benefits of pulp therapy include: removing cavitations or defects to eliminate areas that are susceptible to caries; stopping the progression of tooth demineralization; restoring the integrity of tooth structure; preventing the spread of infection and preventing the shifting of teeth due to loss of tooth structure. The risks of pulp therapy include lessening the longevity of teeth by making them more susceptible to fracture as after removal of gross caries lesion and gaining access to the pulp the tooth become too weak, recurrent lesions, restoration failure, complications, and iatrogenic damage to adjacent teeth.

There are different techniques can be used for gaining intracanal retention in primary teeth. one of these techniques is resin composite posts.

Composite post restorations have been in used in primary teeth from 1986. They yield satisfactory results when there is normal masticatory function, a balanced diet, and hygiene control.

The evidence to support any method of intracanal reinforcement for restoring grossly broken down anterior teeth is presently lacking.

This study aims to Evaluate the intracanal reinforcement with short composite post in upper primary incisors versus no reinforcement.

ELIGIBILITY:
Inclusion Criteria:

* Children Criteria:

  * Medically free.
  * Cooperative patient.
  * Age (3 - 5 years)

Incisors criteria:

• Upper primary incisors show large carious lesions.

Radiographic criteria:

• No evidence of internal/external pathologic root resorption.

Exclusion Criteria:

* • Uncooperative children.

  * Children with systemic disease.
  * Refusal of participation in the study.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Crown success | 1 year
  binary ( presence or abscence of the zircon crown)

SECONDARY OUTCOMES:
Clinically :Gingival health. | 1 year
  * A: No obvious sign of inflammation.
  * B: Mild marginal gingivitis - tissue slightly reddened and edematous.
  * C: Moderate marginal gingivitis - tissue obviously reddened and edematous.
  * D: Sever gingivitis - tissue is very sollowen: spontaneous bleeding.
Radiographic assessment. | 1 year
  * A: Healthy no pathosis noted.
  * B: Pathosis apparent but not requiring immediate treatment.
  * C: Pathosis apparent requiring immediate treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rana T Brtaw, Lecturer, Study Director — Cairo University; Ahmed H Elkadem, professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided